CLINICAL TRIAL: NCT04476524
Title: Clinical and Economic Impact of an Organized Treatment Pathway on Atrial Fibrillation Patient Management From the Emergency Room
Brief Title: Clinical and Economic Impact of an Organized Treatment Pathway on AFib Patient Management From the ER
Acronym: ER2EP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: KCHRF-ER2EP-0004
Record Dates: First submitted 2020-07-14; First posted 2020-07-20 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Cardiac Arrhythmia; Atrial Fibrillation
Keywords: Clinical and Economical impact; Treatment pathway; Emergency Room; Atrial Fibrillation
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation; Emergencies | interventions — Quality Improvement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Arm: Patients who present with AF as the primary diagnosis to the ER will have their chart reviewed
  Interventions: Other: Quality improvement
- Historical Cohort: Historical control arm will be selected from chart review of emergency department prior to the commencement of this study after propensity matching with age and sex.
  Interventions: Other: Quality improvement

INTERVENTIONS:
Other: Quality improvement — All patients with AF as primary problem treated with study protocol would be compared with historical cohort of AF patients who were treated with routine care in the ER. Patients will be followed up and outcomes will be compared between two groups at 1, 3, 6 and 12 months.
  Other Names: All patients with AF as primary problem treated with study protocol would be compared with historical cohort of AF patients who were treated with routine care in the ER.

SUMMARY:
Investigators developed a multidimensional protocol for the management of AF in the emergency department. Investigators aimed to assess if this new ER AF management protocol would result in better outcomes compared to routine care.

DETAILED DESCRIPTION:
Management variation such as selecting rate vs rhythm control, timing and need for thromboembolic treatment, ER vs inpatient treatment and cardiology consultation could lead to disparate care of patients. Therefore, there is a need for future studies to standardize practice leading to improved management, decreased rates of hospitalization and overall cost. Investigators developed a multidimensional protocol for the management of AF in the emergency department. Investigators aimed to assess if this new ER AF management protocol would result in better outcomes compared to routine care.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients > 18 years of age who comes to the ER with AF as the primary diagnosis and is treated according to study protocol.

Exclusion Criteria:

* Patients with established cardiology or electrophysiology care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: i) Study arm: Patients > 18 years of age (both males and females) who present with AF as the primary diagnosis to the ER will have their chart reviewed.
  ii) Historical control arm:Historical control arm will be selected from chart review of emergency department prior to the commencement of this study after propensity matching with age and sex. All patients > 18 years of age (both males and females) who presented with AF as primary diagnosis to the ER of the participating centers within last 2 years will be selected if they meet the inclusion/exclusion criteria mentioned below
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative resource utilization in dollars | 15 months
  Primary Outcome
Time to definitive therapy (AAD and or Ablation) | 15 months
  Primary Outcome
Number of Hospital/clinic visits | 15 months
  Primary Outcome

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, Principal Investigator — Kansas City Heart Rhythm Research Foundation
Locations (1):
- Kansas City Heart Rhythm Institute, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chugh SS, Havmoeller R, Narayanan K, Singh D, Rienstra M, Benjamin EJ, Gillum RF, Kim YH, McAnulty JH Jr, Zheng ZJ, Forouzanfar MH, Naghavi M, Mensah GA, Ezzati M, Murray CJ. Worldwide epidemiology of atrial fibrillation: a Global Burden of Disease 2010 Study. Circulation. 2014 Feb 25;129(8):837-47. doi: 10.1161/CIRCULATIONAHA.113.005119. Epub 2013 Dec 17. PMID 24345399
- [Background] Savelieva I, Camm J. Update on atrial fibrillation: part I. Clin Cardiol. 2008 Feb;31(2):55-62. doi: 10.1002/clc.20138. PMID 18257025
- [Background] Dagres N, Chao TF, Fenelon G, Aguinaga L, Benhayon D, Benjamin EJ, Bunch TJ, Chen LY, Chen SA, Darrieux F, de Paola A, Fauchier L, Goette A, Kalman J, Kalra L, Kim YH, Lane DA, Lip GYH, Lubitz SA, Marquez MF, Potpara T, Pozzer DL, Ruskin JN, Savelieva I, Teo WS, Tse HF, Verma A, Zhang S, Chung MK; ESC Scientific Document Group. European Heart Rhythm Association (EHRA)/Heart Rhythm Society (HRS)/Asia Pacific Heart Rhythm Society (APHRS)/Latin American Heart Rhythm Society (LAHRS) expert consensus on arrhythmias and cognitive function: what is the best practice? Europace. 2018 Sep 1;20(9):1399-1421. doi: 10.1093/europace/euy046. No abstract available. PMID 29562326
- [Background] Tse G, Lip GYH, Liu T. The CHADS2 and CHA2DS2-VASc scores for predicting healthcare utilization and outcomes: Observations on the Appropriate Use and Misuse of Risk scores. Int J Cardiol. 2017 Oct 15;245:181-182. doi: 10.1016/j.ijcard.2017.07.109. No abstract available. PMID 28874290
- [Background] Rozen G, Hosseini SM, Kaadan MI, Biton Y, Heist EK, Vangel M, Mansour MC, Ruskin JN. Emergency Department Visits for Atrial Fibrillation in the United States: Trends in Admission Rates and Economic Burden From 2007 to 2014. J Am Heart Assoc. 2018 Jul 20;7(15):e009024. doi: 10.1161/JAHA.118.009024. PMID 30030215
- [Background] Scheuermeyer FX, Innes G, Pourvali R, Dewitt C, Grafstein E, Heslop C, MacPhee J, Ward J, Heilbron B, McGrath L, Christenson J. Missed opportunities for appropriate anticoagulation among emergency department patients with uncomplicated atrial fibrillation or flutter. Ann Emerg Med. 2013 Dec;62(6):557-565.e2. doi: 10.1016/j.annemergmed.2013.04.004. Epub 2013 May 24. PMID 23711880
- [Background] Funk AM, Kocher KE, Rohde JM, West BT, Crawford TC, Froehlich JB, Saberi S. Variation in practice patterns among specialties in the acute management of atrial fibrillation. BMC Cardiovasc Disord. 2015 Mar 12;15:21. doi: 10.1186/s12872-015-0009-1. PMID 25880061
- [Background] Rogenstein C, Kelly AM, Mason S, Schneider S, Lang E, Clement CM, Stiell IG. An international view of how recent-onset atrial fibrillation is treated in the emergency department. Acad Emerg Med. 2012 Nov;19(11):1255-60. doi: 10.1111/acem.12016. PMID 23167856